CLINICAL TRIAL: NCT00631904
Title: SMDC Pacemaker-MRI Cohort Study
Brief Title: St. Mary's Duluth Clinic (SMDC) Pacemaker Magnetic Resonance Imaging (MRI) Study
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Responsible Party: Michael Mollerus, MD, Essentia Health
Other Study IDs: 010503
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease
Keywords: Pacemaker
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Observation: Patients with permanent pacemakers undergoing medically indicated MRI scanning.

SUMMARY:
The purpose of this study is to monitor and follow non-pacemaker dependent patients with implanted permanent pacemakers, who undergo medically required Magnetic Resonance Imaging (MRI) scans.

Patients with pacemakers are currently excluded from obtaining MRI scans. MRI scanning is now the imaging of choice for a number of neurological, vascular, or musculoskeletal conditions.

Data suggests that patients with pacemakers, when properly monitored, can safely undergo MRI scanning, though the largest published study to date consists of 54 patients, and no long term follow-up has been published.

Though MRI cardiac scanning has been demonstrated to produce local tissue heating at the pacemaker lead tip, the long term effect of tissue heating on lead stability is unclear.

This study will evaluate patients with permanent pacemakers undergoing medically indicated MRI scanning.

Patients will be followed for one year at 3, 6, and 12 months. Data collected will evaluate change in pacing thresholds over time as well as cardiac troponin I, creatinine kinase MB function, and myoglobin levels within the first 12 hours following the scans, side effects, symptoms, the need to make pacemaker program changes, and possible artifacts created by the pacemaker on the MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Permanent pacemaker or ICD implanted for at least 6 weeks
* Referred for medically indicated MRI
* Age greater or equal to 18 years old

Exclusion Criteria:

* ICD market released before 2001 including GDT Ventak-AV, GDT MINI-II, GDT MINI-IV, GDT MINI-III, GDT Prizm-2 MDT GEM-I series
* Epicardial coronary sinus lead or subcutaneous array
* Unable to program all leads to bipolar configuration
* Pacemaker Dependent
* Device has reached elective replacement or end of life
* Other usual contraindications to MRI scanning
* The use of inotropic pharmacological agents, such as dobutamine, during the MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Permanent pacemaker or implantable cardioverter-defibrillator (ICD) implanted for at least 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-01; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Any change greater than 1 volt at a pulse width of 0.5 ms in a pacemaker lead 12 months from an MRI scan | 12 months

SECONDARY OUTCOMES:
Cardiac troponin-I, creatine kinase, MB fraction, and myoglobin levels within the first 12 hours following the scans. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mollerus, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

REFERENCES:
- [Background] Erlebacher JA, Cahill PT, Pannizzo F, Knowles RJ. Effect of magnetic resonance imaging on DDD pacemakers. Am J Cardiol. 1986 Feb 15;57(6):437-40. doi: 10.1016/0002-9149(86)90768-x. PMID 3946261
- [Background] Sommer T, Vahlhaus C, Lauck G, von Smekal A, Reinke M, Hofer U, Block W, Traber F, Schneider C, Gieseke J, Jung W, Schild H. MR imaging and cardiac pacemakers: in-vitro evaluation and in-vivo studies in 51 patients at 0.5 T. Radiology. 2000 Jun;215(3):869-79. doi: 10.1148/radiology.215.3.r00jn08869. PMID 10831713
- [Background] Shellock FG, O'Neil M, Ivans V, Kelly D, O'Connor M, Toay L, Crues JV. Cardiac pacemakers and implantable cardioverter defibrillators are unaffected by operation of an extremity MR imaging system. AJR Am J Roentgenol. 1999 Jan;172(1):165-70. doi: 10.2214/ajr.172.1.9888762.
- [Background] Roguin A, Zviman MM, Meininger GR, Rodrigues ER, Dickfeld TM, Bluemke DA, Lardo A, Berger RD, Calkins H, Halperin HR. Modern pacemaker and implantable cardioverter/defibrillator systems can be magnetic resonance imaging safe: in vitro and in vivo assessment of safety and function at 1.5 T. Circulation. 2004 Aug 3;110(5):475-82. doi: 10.1161/01.CIR.0000137121.28722.33. Epub 2004 Jul 26. PMID 15277324
- [Background] Nazarian S, Roguin A, Zviman MM, Lardo AC, Dickfeld TL, Calkins H, Weiss RG, Berger RD, Bluemke DA, Halperin HR. Clinical utility and safety of a protocol for noncardiac and cardiac magnetic resonance imaging of patients with permanent pacemakers and implantable-cardioverter defibrillators at 1.5 tesla. Circulation. 2006 Sep 19;114(12):1277-84. doi: 10.1161/CIRCULATIONAHA.105.607655. Epub 2006 Sep 11. PMID 16966586
- [Background] Gimbel JR, Bailey SM, Tchou PJ, Ruggieri PM, Wilkoff BL. Strategies for the safe magnetic resonance imaging of pacemaker-dependent patients. Pacing Clin Electrophysiol. 2005 Oct;28(10):1041-6. doi: 10.1111/j.1540-8159.2005.00230.x. PMID 16221260
- [Background] Hayes DL, Holmes DR Jr, Gray JE. Effect of 1.5 tesla nuclear magnetic resonance imaging scanner on implanted permanent pacemakers. J Am Coll Cardiol. 1987 Oct;10(4):782-6. doi: 10.1016/s0735-1097(87)80270-x. PMID 3655146
- [Background] Goldschlager N, Epstein A, Friedman P, Gang E, Krol R, Olshansky B; North American Society of Pacing and Electrophysiology (NASPE) Practice Guideline Committee. Environmental and drug effects on patients with pacemakers and implantable cardioverter/defibrillators: a practical guide to patient treatment. Arch Intern Med. 2001 Mar 12;161(5):649-55. doi: 10.1001/archinte.161.5.649. No abstract available. PMID 11231696
- [Background] Martin ET, Coman JA, Shellock FG, Pulling CC, Fair R, Jenkins K. Magnetic resonance imaging and cardiac pacemaker safety at 1.5-Tesla. J Am Coll Cardiol. 2004 Apr 7;43(7):1315-24. doi: 10.1016/j.jacc.2003.12.016. PMID 15063447
- [Background] Fetter J, Aram G, Holmes DR Jr, Gray JE, Hayes DL. The effects of nuclear magnetic resonance imagers on external and implantable pulse generators. Pacing Clin Electrophysiol. 1984 Jul;7(4):720-7. doi: 10.1111/j.1540-8159.1984.tb05602.x. PMID 6205375